CLINICAL TRIAL: NCT02332421
Title: A Comparison Of The Short-Term Therapeutic Effects Between Two Distractors Used For The Retraction Of Maxillary Canines By Dentoalveolar Distraction Osteogenesis
Brief Title: The Use of a Modified Dentoalveolar Distractor to Retract Maxillary Canines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-OMFS-02-2015
Record Dates: First submitted 2015-01-03; First posted 2015-01-06 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-01

CONDITIONS: Orthodontic Patients Requiring Canine Retraction
Keywords: canine retraction; acceleration of tooth movement; dentoalveolar distraction osteogenesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- modified dentoalveolar distractor (Experimental): Canine retraction will be accomplished using a modified dentoalveolar distractor
  Interventions: Device: modified dentoalveolar distractor
- conventional dentoalveolar distractor (No Intervention): Canine retraction will be accomplished using a conventional dentoalveolar distractor

INTERVENTIONS:
Device: modified dentoalveolar distractor — Here, the modified distractor is going to be used when retracting the canine.
  Arms: modified dentoalveolar distractor

SUMMARY:
In this study, two distractors will be used to retract maxillary canines into the extraction sites. The first distractor is a modified Hyrax expander with two arms soldered to two bands connected to a canine and a molar; and the second one is a similar to the first one but with the addition of a third arm.

The purpose of this investigation is to compare the two distractors in terms of: final position of the canine, canine pulp vitality, molars' anchorage, patient's acceptance to the appliance.

DETAILED DESCRIPTION:
The retraction of the canines is one of the longest and most important stages in the orthodontic treatment of cases that require premolars extraction. The retraction phase of the canines into an extraction site with conventional treatment method usually lasts about 4 to 6 months under normal circumstances. The use of dentoalveolar distraction (DAD) technique has been considered a very important step in this field. It has been shown by early case reports that this technique can be employed to retract canines within 10 to 14 days.

Although DAD is thought to accelerate tooth movement during canine retraction, a significant amount of tipping (distal tilting) was observed in many case reports. So in this study, there is an intention to apply a modified DAD device on one side of the mouth and to compare it with the conventional one applied on the opposite side of the mouth in each participating patient.

ELIGIBILITY:
Inclusion Criteria:

* Indication for extraction of upper first premolar and conducting canine retraction
* Good oral hygiene

Exclusion Criteria:

* Buccal or palatal inclination of the canines
* Mesial or distal inclination of the canines
* Contraindication to minor surgery
* Previous orthodontic or surgical treatment
* Root canal treatment to the canines
* Malformation of the canines

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in the mesiodistal inclination of the canine | This will be measured at three times: T0, one day before installing the distractor; T1, in the same day of finishing the retraction phase; T2, in the same day of device removal from the mouth.
  This will be measured using a lateral cephalogram taken at these assessment times. The long axis of the canine will be drawn on the tracing of the cephalogram at each assessment time and this long axis will be measured with reference to anterior cranial base.

SECONDARY OUTCOMES:
Change in Canine Pulp Vitality | This will be measured at three times: T0, one day before installing the distractor; T1, in the same day of finishing the retraction phase; T2, in the same day of device removal from the mouth.
  This variable is going to be measured clinically
Molars Anchorage Loss | Upper first molar position will be measured at three assessment times: T0, one day before installing the distractor; T1, in the same day of finishing the retraction phase; T2, in the same day of device removal from the mouth.
  This will be measured using cephalograms and study models
Patient acceptance to each distractor | This is going to be measured at: (T1) first day following surgery, (T2) five days following surgery, (T3) two weeks following surgery, and (T4) at the time of appliance removal.
  Using a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Alainawi, DDS, Principal Investigator — MSc student, Oral and Maxillofacial Surgery Department, University of Damascus Dental School; Yassir Al-Medallal, DDS MSc PhD, Study Director — Associate Professor of Oral and Maxillofacial Surgery, University of Damascus Dental School; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor of Orthodontics, University of Damascus Dental School
Locations (1):
- Department of Oral and Maxillofacial Surgery, University of Damascus Dental School, Damascus, Damscus, Syria

REFERENCES:
- [Background] Kurt G, Iseri H, Kisnisci R. Rapid tooth movement and orthodontic treatment using dentoalveolar distraction (DAD). Long-term (5 years) follow-up of a Class II case. Angle Orthod. 2010 May;80(3):597-606. doi: 10.2319/041209-209.1. PMID 20050758
- [Background] Sukurica Y, Karaman A, Gurel HG, Dolanmaz D. Rapid canine distalization through segmental alveolar distraction osteogenesis. Angle Orthod. 2007 Mar;77(2):226-36. doi: 10.2319/0003-3219(2007)077[0226:RCDTSA]2.0.CO;2. PMID 17319756
- [Background] Gurgan CA, Iseri H, Kisnisci R. Alterations in gingival dimensions following rapid canine retraction using dentoalveolar distraction osteogenesis. Eur J Orthod. 2005 Aug;27(4):324-32. doi: 10.1093/ejo/cji011. PMID 16043471
- [Background] Kisnisci RS, Iseri H, Tuz HH, Altug AT. Dentoalveolar distraction osteogenesis for rapid orthodontic canine retraction. J Oral Maxillofac Surg. 2002 Apr;60(4):389-94. doi: 10.1053/joms.2002.31226. PMID 11928095
- [Background] Nair A, Kumar JP, Venkataramana V, Yuvaraj A, Reddy VS, Kumar SK. Dento-Alveolar distraction osteogenesis using rigid intra-oral tooth borne distraction device. J Int Oral Health. 2014 Apr;6(2):106-13. Epub 2014 Apr 26. PMID 24876710
- [Background] Kumar N, Prashantha G, Raikar S, Ranganath K, Mathew S, Nambiar S. Dento-Alveolar Distraction Osteogenesis for rapid Orthodontic Canine Retraction. J Int Oral Health. 2013 Dec;5(6):31-41. Epub 2013 Dec 26. PMID 24453442